CLINICAL TRIAL: NCT03336073
Title: Carfilzomib and Dexamethasone in Combination With Cyclophosphamide vs. Carfilzomib and Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma: a Phase II Randomized Controlled Trial
Brief Title: Carfilzomib, Cyclophosphamide, Dexamethasone in Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM-KyCyDex
Record Dates: First submitted 2017-10-25; First posted 2017-11-08 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carfilzomib, dexamethasone and cyclophosphamide (Experimental): carfilzomib at a dose of 70 mg/m2 (20 mg/m2 only in the first infusion) intravenously (iv) on days 1, 8, and 15, dexamethasone by mouth (po) at a dose of 20 mg (10 mg for patients >75 years) days 1, 2, 8, 9, 15 and 16 and cyclophosphamide at a dose of 300 mg/m2 iv on days 1, 8 and 15, in 28 days cycles
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: cyclophosphamide
- carfilzomib and dexamethasone (Active Comparator): carfilzomib at a dose of 70 mg/m2 (20 mg/m2 only in the first infusion) intravenously (iv) on days 1, 8, and 15, dexamethasone by mouth (po) at a dose of 20 mg (10 mg for patients >75 years) days 1, 2, 8, 9, 15 and 16 , in 28 days cycles
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — carfilzomib at a dose of 70 mg/m2 (20 mg/m2 only in the first infusion) intravenously (iv) on days 1, 8, and 15
Drug: Dexamethasone — dexamethasone oral at a dose of 20 mg (10 mg for patients >75 years) days 1, 2, 8, 9, 15 and 16
Drug: cyclophosphamide — cyclophosphamide at a dose of 300 mg/m2 iv on days 1, 8 and 15
  Arms: carfilzomib, dexamethasone and cyclophosphamide

SUMMARY:
This is a multicenter, open label, phase II randomized controlled study that will evaluate the efficacy of carfilzomib and dexamethasone in combination with cyclophosphamide in R/R MM patients.

For this purpose, R/R MM patients that have received 1-3 prior lines of therapy, and who are not primary refractory or refractory to proteasome inhibitors will be randomized to receive:

* Experimental arm: carfilzomib at a dose of 70 mg/m2 (20 mg/m2 only in the first infusion) intravenously (iv) on days 1, 8, and 15, dexamethasone by mouth (po) at a dose of 20 mg (10 mg for patients >75 years) days 1, 2, 8, 9, 15 and 16 and cyclophosphamide at a dose of 300 mg/m2 iv on days 1, 8 and 15, in 28 days cycles; or
* Control arm: the same treatment but without cyclophosphamide.

Once the first 12 cycles are administered, treatment will be administered on days 1 and 15 of each cycle and the visit and doses on day 8 will be omitted in both study arms.

Patients older than 75 years will receive in both arms carfilzomib at a dose of 56 mg/m2 (20 mg/m2 only in the first infusion) during the cycles 1 and 2. If tolerability is acceptable, the dose could be increased up to 70 mg/m2 since the cycle 3.

Treatment will be continued until progression, unacceptable toxicity or investigator or patient decision.

DETAILED DESCRIPTION:
Treatment will consist of 28-days cycles with:

* Arm 1 (experimental arm):

  * Carfilzomib administered iv at a dose of 70 mg/m2 (20 mg/m2 only in the first infusion) iv on days 1, 8 and 15.
  * Dexamethasone at a dose of 20 mg po (10 mg for patients >75 years) days 1, 2, 8, 9, 15 and 16.
  * Cyclophosphamide at a dose of 300 mg/m2 iv on days 1, 8 and 15
* Arm 2 (control arm):

  * Carfilzomib administered iv at a dose of 70 mg/m2 (20 mg/m2 only in the first infusion) iv on days 1, 8, and 15.
  * Dexamethasone at a dose of 20 mg po (10 mg for patients >75 years) days 1, 2, 8, 9, 15 and 16.

Once the first 12 cycles are administered, treatment will be administered on days 1 and 15 of each cycle and the visit and doses on day 8 will be omitted in both study arms.

Patients older than 75 years will receive in both arms carfilzomib at a dose of 56 mg/m2 (20 mg/m2 only in the first infusion) during the cycles 1 and 2. If tolerability is acceptable, the dose could be increased up to 70 mg/m2 since the cycle 3.

Treatments will be administered until progressive disease (PD) or unacceptable toxicity. Carfilzomib and cyclophosphamide will be provided by the sponsor. Dexamethasone may be utilized per a site's standard practice and will not be provided by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Performance status (ECOG) <2.
3. Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
4. Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
5. Patients previously diagnosed with MM according to the IMWG criteria (Lancet Oncology 2014) that after previous treatment with 1-3 regimens require therapy due to a relapse/progression of the disease.
6. Patients must have measurable disease, defined as follows:

   * Serum monoclonal protein ≥ 0.5 g/L, or
   * Urine light-chain excretion of ≥ 0.2g /24 hours, or
   * Abnormal ratio of serum free light chains (FLCs) plus involved FLC level ≥100 mg/L.

Exclusion Criteria:

1. Primary refractory patients defined as not having achieved at least a PR with a prior therapy.
2. Refractoriness to prior proteasome inhibitor therapies, defined as not having achieved at least MR or having progressed under treatment or in the first 60 days after the last dose of the proteasome inhibitor.
3. Biochemical and haematological abnormalities as specified below:

   * Hemoglobin < 8.0 g/dL.
   * Platelet count <75x109/L without previous platelet transfusions in the last 7 days. If bone marrow infiltration is greater than 50%, a platelet count of ≥50x109/L is required.
   * Absolute neutrophil count (ANC) < 0.75 x109/L without G-CSF support in the last 7 days.
   * Aspartate transaminase (AST): > 2.5 times the upper limit of normal.
   * Alanine transaminase (ALT): > 2.5 times the upper limit of normal.
   * Calculated or measured creatinine clearance: <30 mL/min (calculated from the Cockcroft and Gault formula, specified in Appendix C).
4. Left ventricle ejection fraction < 50%.
5. Absence of recovery from any significant non-haematological toxicity derived from previous treatments. The presence of alopecia and NCI-CTC grade < 2 symptomatic peripheral neuropathy is allowed.
6. Pregnant or breastfeeding women; men and women of reproductive potential who are not using effective contraceptive methods (double barrier method, intrauterine device, and oral contraception).
7. Previous history of any other neoplastic disease in the last five years (except basal cell carcinoma, skin epithelioma or carcinoma in situ of any site).
8. Other relevant diseases or adverse clinical conditions:

   * Congestive heart failure or angina pectoris, myocardial infarction within 12 months before inclusion in the study.
   * Uncontrolled arterial hypertension or cardiac arrhythmias (i.e. requiring a change in medication within the last 3 months or a hospital admission within the past 6 months).
   * History of significant neurological or psychiatric disorders.
   * Active infection
   * Significant non-neoplastic liver disease (e.g. cirrhosis, active chronic hepatitis).
9. Patient is known to be human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive or to suffer active hepatitis C infection
10. The patient has received concomitant anti-myeloma therapy within 14 days prior to Day 1 of Cycle 1.
11. Limit to the patient's ability to comply with the treatment or follow-up protocol.
12. Uncontrolled endocrine diseases (e.g. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 36 months
  PFS is defined as the number of months from randomization to the disease progression or death due to any cause, whichever occurs first. The disease outcome determined will be the primary data source for the final PFS analysis.

SECONDARY OUTCOMES:
Safety of carfilzomib, dexamethasone and cyclophosphamide in number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  the safety as determined by the incidence of clinical and laboratory toxicities
Efficacy of carfilzomib, dexamethasone and cyclophosphamide in number and rate of responses obtained | 2 years
  Evaluate the efficacy of carfilzomib and dexamethasone in combination with cyclophosphamide in terms of rate of response in multiple myeloma (MM) patients.
Time-to progression (TTP) | 36 months
  Duration from randomization to disease progression, with deaths due to causes other than progression censored.
Overall Survival (OS) | 36 months
  Duration from the date of randomization until the date of death. The patients lost to follow-up will be censored at the date of the last visit.
Efficacy of carfilzomib, dexamethasone and cyclophosphamide in rate of achievement of immunophenotypic CR | 2 years
  Evaluate the efficacy of carfilzomib and dexamethasone in combination with cyclophosphamide in terms of achievement of immunophenotypic CR in multiple myeloma (MM) patients.

CONTACTS AND LOCATIONS:
Locations (24):
- Spain (24):
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - H.Universitari Germans Trias I Pujol de Badalona, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Ico L'Hospitalet, Barcelona
  - Complejo Hospitalario de Cáceres, Cáceres
  - Hospital de Cabueñes, Gijón
  - Centro Hospitalario Universitario de Granada, Granada
  - Hospital de León, León
  - H. 12 de Octubre, Madrid
  - H. Ramón y Cajal, Madrid
  - Hospital Sanchinarro, Madrid
  - Hospital Costa del Sol, Málaga
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Virgn de la Arrixaca, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital de Son Llàtzer, Palma de Mallorca
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario de Santiago, Santiago de Compostela
  - Hospital de Segovia, Segovia
  - Complejo Hospitalario Regional Virgen Del Rocío, Seville
  - Hospital de Toledo, Toledo
  - Hospital Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Cancer Society. Cancer facts and figures 2005. Atlanta, GA: American Cancer Society 2005.
- [Background] Arastu-Kapur S, Shenk K, Kirk CJ, et al. Nonproteasomal targets of proteasome inhibitors bortezomib and carfilzomib. Haematologica. 2009:94(s2). 14th Congress of the European Hematology Association 2009. Abstract 0939.
- [Background] Berenson JR, Cartmell A, Bessudo A, Lyons RM, Harb W, Tzachanis D, Agajanian R, Boccia R, Coleman M, Moss RA, Rifkin RM, Patel P, Dixon S, Ou Y, Anderl J, Aggarwal S, Berdeja JG. CHAMPION-1: a phase 1/2 study of once-weekly carfilzomib and dexamethasone for relapsed or refractory multiple myeloma. Blood. 2016 Jun 30;127(26):3360-8. doi: 10.1182/blood-2015-11-683854. Epub 2016 May 12. PMID 27207788
- [Background] Boyle P, Ferlay J. Cancer incidence and mortality in Europe, 2004. Ann Oncol. 2005 Mar;16(3):481-8. doi: 10.1093/annonc/mdi098. Epub 2005 Feb 17. PMID 15718248
- [Background] Bringhen S, Petrucci MT, Larocca A, Conticello C, Rossi D, Magarotto V, Musto P, Boccadifuoco L, Offidani M, Omede P, Gentilini F, Ciccone G, Benevolo G, Genuardi M, Montefusco V, Oliva S, Caravita T, Tacchetti P, Boccadoro M, Sonneveld P, Palumbo A. Carfilzomib, cyclophosphamide, and dexamethasone in patients with newly diagnosed multiple myeloma: a multicenter, phase 2 study. Blood. 2014 Jul 3;124(1):63-9. doi: 10.1182/blood-2014-03-563759. Epub 2014 May 22. PMID 24855212
- [Background] Demo SD, Kirk CJ, Aujay MA, Buchholz TJ, Dajee M, Ho MN, Jiang J, Laidig GJ, Lewis ER, Parlati F, Shenk KD, Smyth MS, Sun CM, Vallone MK, Woo TM, Molineaux CJ, Bennett MK. Antitumor activity of PR-171, a novel irreversible inhibitor of the proteasome. Cancer Res. 2007 Jul 1;67(13):6383-91. doi: 10.1158/0008-5472.CAN-06-4086. PMID 17616698
- [Background] de Waal EG, de Munck L, Hoogendoorn M, Woolthuis G, van der Velden A, Tromp Y, Vellenga E, Hovenga S. Combination therapy with bortezomib, continuous low-dose cyclophosphamide and dexamethasone followed by one year of maintenance treatment for relapsed multiple myeloma patients. Br J Haematol. 2015 Dec;171(5):720-5. doi: 10.1111/bjh.13653. Epub 2015 Sep 11. PMID 26358087
- [Background] Dimopoulos MA, Moreau P, Palumbo A, Joshua D, Pour L, Hajek R, Facon T, Ludwig H, Oriol A, Goldschmidt H, Rosinol L, Straub J, Suvorov A, Araujo C, Rimashevskaya E, Pika T, Gaidano G, Weisel K, Goranova-Marinova V, Schwarer A, Minuk L, Masszi T, Karamanesht I, Offidani M, Hungria V, Spencer A, Orlowski RZ, Gillenwater HH, Mohamed N, Feng S, Chng WJ; ENDEAVOR Investigators. Carfilzomib and dexamethasone versus bortezomib and dexamethasone for patients with relapsed or refractory multiple myeloma (ENDEAVOR): a randomised, phase 3, open-label, multicentre study. Lancet Oncol. 2016 Jan;17(1):27-38. doi: 10.1016/S1470-2045(15)00464-7. Epub 2015 Dec 5. PMID 26671818
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Background] Fu W, Delasalle K, Wang J, Song S, Hou J, Alexanian R, Wang M. Bortezomib-cyclophosphamide-dexamethasone for relapsing multiple myeloma. Am J Clin Oncol. 2012 Dec;35(6):562-5. doi: 10.1097/COC.0b013e31822043f6. PMID 21694573
- [Background] Garcia-Sanz R, Gonzalez-Porras JR, Hernandez JM, Polo-Zarzuela M, Sureda A, Barrenetxea C, Palomera L, Lopez R, Grande-Garcia C, Alegre A, Vargas-Pabon M, Gutierrez ON, Rodriguez JA, San Miguel JF. The oral combination of thalidomide, cyclophosphamide and dexamethasone (ThaCyDex) is effective in relapsed/refractory multiple myeloma. Leukemia. 2004 Apr;18(4):856-63. doi: 10.1038/sj.leu.2403322. PMID 14973508
- [Background] Jawed I, Lee CM, Tward JD, et al. Survival outcomes for multiple myeloma over three decades: A Surveillance, Epidemiology, and End Results (SEER) analysis. J Clin Oncol. 2007;25(18_suppl). ASCO Annual Meeting 2007. Abstract 8019.
- [Background] Kim YK, Sohn SK, Lee JH, Yang DH, Moon JH, Ahn JS, Kim HJ, Lee JJ; Korean Multiple Myeloma Working Party (KMMWP). Clinical efficacy of a bortezomib, cyclophosphamide, thalidomide, and dexamethasone (Vel-CTD) regimen in patients with relapsed or refractory multiple myeloma: a phase II study. Ann Hematol. 2010 May;89(5):475-82. doi: 10.1007/s00277-009-0856-x. Epub 2009 Nov 18. PMID 19921192
- [Background] Kuhn DJ, Chen Q, Voorhees PM, Strader JS, Shenk KD, Sun CM, Demo SD, Bennett MK, van Leeuwen FW, Chanan-Khan AA, Orlowski RZ. Potent activity of carfilzomib, a novel, irreversible inhibitor of the ubiquitin-proteasome pathway, against preclinical models of multiple myeloma. Blood. 2007 Nov 1;110(9):3281-90. doi: 10.1182/blood-2007-01-065888. Epub 2007 Jun 25. PMID 17591945
- [Background] Kumar S, Flinn I, Richardson PG, Hari P, Callander N, Noga SJ, Stewart AK, Turturro F, Rifkin R, Wolf J, Estevam J, Mulligan G, Shi H, Webb IJ, Rajkumar SV. Randomized, multicenter, phase 2 study (EVOLUTION) of combinations of bortezomib, dexamethasone, cyclophosphamide, and lenalidomide in previously untreated multiple myeloma. Blood. 2012 May 10;119(19):4375-82. doi: 10.1182/blood-2011-11-395749. Epub 2012 Mar 15. PMID 22422823
- [Background] Lee SJ, Levitsky K, Parlati F, Bennett MK, Arastu-Kapur S, Kellerman L, Woo TF, Wong AF, Papadopoulos KP, Niesvizky R, Badros AZ, Vij R, Jagannath S, Siegel D, Wang M, Ahmann GJ, Kirk CJ. Clinical activity of carfilzomib correlates with inhibition of multiple proteasome subunits: application of a novel pharmacodynamic assay. Br J Haematol. 2016 Jun;173(6):884-95. doi: 10.1111/bjh.14014. Epub 2016 Apr 12. PMID 27071340
- [Background] Millennium Pharmaceuticals, Inc. Velcade (bortezomib) full prescribing information [package insert]; 2012
- [Background] Morgan GJ, Davies FE, Gregory WM, Russell NH, Bell SE, Szubert AJ, Navarro Coy N, Cook G, Feyler S, Byrne JL, Roddie H, Rudin C, Drayson MT, Owen RG, Ross FM, Jackson GH, Child JA; NCRI Haematological Oncology Study Group. Cyclophosphamide, thalidomide, and dexamethasone (CTD) as initial therapy for patients with multiple myeloma unsuitable for autologous transplantation. Blood. 2011 Aug 4;118(5):1231-8. doi: 10.1182/blood-2011-02-338665. Epub 2011 Jun 7. PMID 21652683
- [Background] Muchtar E, Gertz MA, Magen H. A practical review on carfilzomib in multiple myeloma. Eur J Haematol. 2016 Jun;96(6):564-77. doi: 10.1111/ejh.12749. Epub 2016 Mar 9. PMID 26893241
- [Background] Nijhof IS, Franssen LE, Levin MD, Bos GMJ, Broijl A, Klein SK, Koene HR, Bloem AC, Beeker A, Faber LM, van der Spek E, Ypma PF, Raymakers R, van Spronsen DJ, Westerweel PE, Oostvogels R, van Velzen J, van Kessel B, Mutis T, Sonneveld P, Zweegman S, Lokhorst HM, van de Donk NWCJ. Phase 1/2 study of lenalidomide combined with low-dose cyclophosphamide and prednisone in lenalidomide-refractory multiple myeloma. Blood. 2016 Nov 10;128(19):2297-2306. doi: 10.1182/blood-2016-07-729236. Epub 2016 Sep 19. PMID 27647864
- [Background] O'Connor OA, Stewart AK, Vallone M, Molineaux CJ, Kunkel LA, Gerecitano JF, Orlowski RZ. A phase 1 dose escalation study of the safety and pharmacokinetics of the novel proteasome inhibitor carfilzomib (PR-171) in patients with hematologic malignancies. Clin Cancer Res. 2009 Nov 15;15(22):7085-91. doi: 10.1158/1078-0432.CCR-09-0822. Epub 2009 Nov 10. PMID 19903785
- [Background] Papadopoulos KP, Siegel DS, Vesole DH, Lee P, Rosen ST, Zojwalla N, Holahan JR, Lee S, Wang Z, Badros A. Phase I study of 30-minute infusion of carfilzomib as single agent or in combination with low-dose dexamethasone in patients with relapsed and/or refractory multiple myeloma. J Clin Oncol. 2015 Mar 1;33(7):732-9. doi: 10.1200/JCO.2013.52.3522. Epub 2014 Sep 15. PMID 25225420
- [Background] Reece DE, Masih-Khan E, Atenafu EG, Jimenez-Zepeda VH, Anglin P, Chen C, Kukreti V, Mikhael JR, Trudel S. Phase I-II trial of oral cyclophosphamide, prednisone and lenalidomide for the treatment of patients with relapsed and refractory multiple myeloma. Br J Haematol. 2015 Jan;168(1):46-54. doi: 10.1111/bjh.13100. Epub 2014 Aug 22. PMID 25146584
- [Background] Siegel DS, Martin T, Wang M, Vij R, Jakubowiak AJ, Lonial S, Trudel S, Kukreti V, Bahlis N, Alsina M, Chanan-Khan A, Buadi F, Reu FJ, Somlo G, Zonder J, Song K, Stewart AK, Stadtmauer E, Kunkel L, Wear S, Wong AF, Orlowski RZ, Jagannath S. A phase 2 study of single-agent carfilzomib (PX-171-003-A1) in patients with relapsed and refractory multiple myeloma. Blood. 2012 Oct 4;120(14):2817-25. doi: 10.1182/blood-2012-05-425934. Epub 2012 Jul 25. PMID 22833546
- [Background] Smith TJ, Khatcheressian J, Lyman GH, Ozer H, Armitage JO, Balducci L, Bennett CL, Cantor SB, Crawford J, Cross SJ, Demetri G, Desch CE, Pizzo PA, Schiffer CA, Schwartzberg L, Somerfield MR, Somlo G, Wade JC, Wade JL, Winn RJ, Wozniak AJ, Wolff AC. 2006 update of recommendations for the use of white blood cell growth factors: an evidence-based clinical practice guideline. J Clin Oncol. 2006 Jul 1;24(19):3187-205. doi: 10.1200/JCO.2006.06.4451. Epub 2006 May 8. PMID 16682719
- [Background] Stewart AK, Rajkumar SV, Dimopoulos MA, Masszi T, Spicka I, Oriol A, Hajek R, Rosinol L, Siegel DS, Mihaylov GG, Goranova-Marinova V, Rajnics P, Suvorov A, Niesvizky R, Jakubowiak AJ, San-Miguel JF, Ludwig H, Wang M, Maisnar V, Minarik J, Bensinger WI, Mateos MV, Ben-Yehuda D, Kukreti V, Zojwalla N, Tonda ME, Yang X, Xing B, Moreau P, Palumbo A; ASPIRE Investigators. Carfilzomib, lenalidomide, and dexamethasone for relapsed multiple myeloma. N Engl J Med. 2015 Jan 8;372(2):142-52. doi: 10.1056/NEJMoa1411321. Epub 2014 Dec 6. PMID 25482145
- [Background] Suzuki E, Demo S, Deu E, Keats J, Arastu-Kapur S, Bergsagel PL, Bennett MK, Kirk CJ. Molecular mechanisms of bortezomib resistant adenocarcinoma cells. PLoS One. 2011;6(12):e27996. doi: 10.1371/journal.pone.0027996. Epub 2011 Dec 22. PMID 22216088
- [Background] Vij R, Wang M, Kaufman JL, Lonial S, Jakubowiak AJ, Stewart AK, Kukreti V, Jagannath S, McDonagh KT, Alsina M, Bahlis NJ, Reu FJ, Gabrail NY, Belch A, Matous JV, Lee P, Rosen P, Sebag M, Vesole DH, Kunkel LA, Wear SM, Wong AF, Orlowski RZ, Siegel DS. An open-label, single-arm, phase 2 (PX-171-004) study of single-agent carfilzomib in bortezomib-naive patients with relapsed and/or refractory multiple myeloma. Blood. 2012 Jun 14;119(24):5661-70. doi: 10.1182/blood-2012-03-414359. Epub 2012 May 3. PMID 22555973
- [Derived] Puertas B, Gonzalez-Calle V, Sureda A, Moreno MJ, Oriol A, Gonzalez E, Rosinol L, Lopez J, Escalante F, Martinez-Lopez J, Carrillo E, Clavero E, Rios-Tamayo R, Rey-Bua B, Gonzalez-Rodriguez AP, Dourdil V, De Arriba F, Gonzalez S, Perez-de-Oteyza J, Hernandez MT, Garcia-Mateo A, Bargay J, Blade J, Lahuerta JJ, San Miguel JF, Ocio EM, Mateos MV. Randomized phase II study of weekly carfilzomib 70 mg/m2 and dexamethasone with or without cyclophosphamide in relapsed and/or refractory multiple myeloma patients. Haematologica. 2023 Oct 1;108(10):2753-2763. doi: 10.3324/haematol.2022.282490. PMID 37102598